# Project Plan Cover Page

# Official Study Title:

Empowering Narratives: Aid to Self-help for Ukrainian Refugees A Randomized Controlled Trial of Narrative Exposure Therapy (NET) Delivered by Supervised Ukrainian Health Professionals in Norway

# ClinicalTrials.gov Identifier (NCT Number):

NCT07062042NCT000000000 (Replace with actual number once registered)

# **Document Type:**

Project Plan – focused on methodological procedures

# Responsible Institution:

Kristiania University College School of Health Sciences and School of Art, Design, and Media

# Principal Investigator:

Vanessa Nolasco Ferreira, PhD Associate Professor, Clinical Psychologist Kristiania University College vanessanolasco.ferreira@kristiania.no

# **Date of Document:**

14th October 2024 12th August 2025

Formatted: Superscript

# Project Plan - methodological procedures

#### Oversight:

Human Subjects Review: REK ref nr. 790305

Board Name: REK sør-øst

Board Affiliation: REK sør-øst A

Phone:+47 22857547

Email: rek-sorost@medisin.uio.no

Address: Gullhaugveien 1-3, 0484 Oslo

#### **Study Description:**

#### **Brief Summary:**

**Background:** The Russian invasion of Ukraine has resulted in forced displacement, with over 80,000 Ukrainian refugees now residing in Norway(1). This displacement, and, in many cases, preceding war experiences, has led to increased vulnerability to trauma and mental health challenges. Narrative Exposure Therapy (NET), a short-term traumafocused intervention, has demonstrated efficacy in reducing PTSD symptoms among individuals exposed to organized violence and war. (2)

**Aim:** The protocol aims to assess the clinical effects of Narrative Exposure Therapy (NET) on PTSD and depression symptoms among Ukrainian refugees in Norway and to facilitate training and supervised praxis for Ukrainian health professionals in using NET.

**Methods**: This study employs a pretest-posttest randomized controlled experimental design. Ukrainian health professionals in Norway will receive standardized NET training through a digital course. Subsequently, they will treat Ukrainian refugees using NET under supervision. Participants will be screened and assessed at three time points: baseline, immediately after treatment, and at 6-month follow-up. Validated instruments in Ukrainian and Russian will be used to assess trauma experiences, symptoms, comorbidities: PHQ-9(3), ITQ(4), LEC-5(5, 6), SHUT-D(7), and demographic questionnaire. Exclusion criteria include active psychotic spectrum disorders, neurodevelopmental disorders and concurrent trauma therapy.

**Ethics and Dissemination**: Ethical approval was sought from REK under the reference number 790305 and SIKT, under the reference number 116071. All data will be anonymized and stored using Services for sensitive data (TSD). Results will be

disseminated through peer-reviewed publications, public presentations, and digital media. Emergency procedures for participants presenting severe mental health symptoms are in place, including psychoeducational consultations and referral to public health services.

#### **Detailed Description:**

#### Background:

The Russian Federation's annexation of Crimea in 2014 marked the beginning of the Russo-Ukrainian conflict. The full-scale invasion launched on February 24, 2022, precipitated a humanitarian crisis, resulting in the largest refugee movement in Europe since World War II. By April 2025, over 6.9 million Ukrainian refugees were recorded globally, with approximately 6.3 million residing in Europe. Norway, with a population of 5.5 million, has been impacted by this influx. As of early 2025, approximately 80 thousand Ukrainian refugees had sought protection in Norway, making Ukrainians the second-largest immigrant group in the country (1)

Epidemiological studies have begun to assess the health status of Ukrainian refugees in Norway analyzing trends in self-reported health among Ukrainian refugees, revealing variations based on the month of arrival in 2022. One study indicated that refugees who arrived later in 2022 generally reported poorer long-term health but less psychological distress than those who arrived earlier in the year(8). In what concerns mental health, an assessment of the self-reported health status and healthcare needs of Ukrainian refugees who arrived in Norway in 2022 showed that the mean score on the Hopkins Symptom Checklist (HSCL-5) was 2.24 among Ukrainian refugees, indicating higher psychological distress compared to the Norwegian average of 1.60(9).

Although some research has been conducted no studies, to our knowledge, have examined effects of structured mental health interventions for Ukrainian refugees in Norway. This study will evaluate the use of Narrative Exposure Therapy (NET) to address trauma-related symptoms among Ukrainian Adults that have sought collective protection in Norway after February 2022.

Narrative Exposure Therapy (NET) is a short-term, trauma-focused intervention developed for individuals exposed to multiple traumatic events, including refugees and survivors of war and organized violence. It is grounded in principles of cognitive-behavioral therapy and testimonial therapy. NET helps adults reconstruct a coherent narrative of their life by integrating fragmented traumatic memories through structured exposure within a chronological autobiographical framework. Core components include lifeline construction, imaginal exposure to traumatic events, and reprocessing of emotional responses. The method emphasizes stabilization through therapeutic structure and is supported by evidence from randomized controlled trials showing

reductions in PTSD symptoms. The approach is protocol-driven and applicable in low-resource settings under supervision, as outlined in the practice document.

The study also involves training Ukrainian health workers and professionals in Norway to deliver NET, with the goal of assessing outcomes and examining how such an approach can be implemented within refugee communities.

#### Objectives:

- To evaluate the effect of NET on PTSD, depression and dissociation symptoms among Ukrainian refugees in Norway.
- To train Ukrainian health professionals in Norway to deliver NET and facilitate their professional integration.
- To collect longitudinal data on trauma symptomatology and treatment outcomes.

#### Structure - Training Health Workers

The training program conducted from January 6th to 17th consisted of a total of 1,755 minutes, which equals 29 hours and 15 minutes of structured education and practice. The curriculum covered a comprehensive range of topics relevant to trauma-informed care and Narrative Exposure Therapy (NET). Key areas addressed included foundational knowledge on violence, PTSD, and dissociation (with references to WHO and ICD-11), as well as the role of shame and guilt in trauma. Ethical and relational aspects were highlighted through sessions on therapeutic alliance and Norwegian ethical guidelines. Technical and clinical skills were developed through lectures and hands-on practice related to mental health screening, the lifeline method, and NET's core techniques, including processing of traumatic and positive memories ("stones," "sticks," and "flowers"). Further content addressed FORNET and rapid NET, NETfacts, and psychohygiene. The training combined theory-based lectures with practical small group exercises to support participants in applying NET principles in real-world settings. In addition to the training, a total of 51 group supervision sessions of 90 minutes each, involving 6 health professionals and workers per supervision were offered to the 21 health workers in the project. Each of them must prepare and present the case progression in at least 10 supervision sessions. Two health workers / professionals present per supervision session and the other 4 discuss the case with guidance of a supervisor that has a psychologist or a psychiatrist background.

To ensure adherence to the NET Manual some fidelity measures were included. All the health workers receive a hands-on material in Ukrainian with the content and instructions for each step of the treatment (screening, lifeline session, exposure sessions, and final session with the re-reading of the participant's whole narrative). A

Formatted: Font: Not Bold

check list with the course and order of the sessions are also provided to ensure that the study design will be followed. As self-report measures the health workers, after every session, must, in maximum 24 hours, report through a specific form (Nettskjema) the content of the sessions and any difficulties, disturbances, request of the participant that are under treatment, and the use of any different approach that were not predict in the guidelines. The form is connected directly to a security system (TSD), complying with all the GDPR regulations and ethical requirements, forming a participant journal. The primary investigator and the supervisors access the journals and advise the health workers ensuring that the premises of NET and the design of the study are being followed, this is part of the assessor report measures, that also include rating the percentage that each health work adhered to the NET manual and followed the instructions provided.

#### Study Design and Methodology

#### Design:

This is a pretest-posttest randomized controlled experimental study with two arms: immediate treatment group and wait-list control group. The intervention consists of 8–12 NET sessions delivered individually, depending on the number of sessions each participant needs in order to create a coherent story of their life and depending on the number of traumatic experiences reported in the LEC5.

## **Participants and Recruitment**

Participants include Ukrainian refugees aged 18+, residing in Norway, with trauma exposure related to war or forced displacement. Ukrainian health professionals will recruit patients via community outreach and referrals. Every health professional will be assigned to participants based on their place of residence in order to minimize travel time to therapy sessions. Within each pair of participants, the allocation to treatment group and wait-list control group will be random sorted in Excel.

## **Inclusion and Exclusion Criteria**

Inclusion: Ukrainian adult refugees, exposure to war or flight trauma, and informed consent.

Exclusion: Active psychotic symptoms, neurodevelopmental disorders, concurrent trauma therapy, or severe cognitive impairment.

## Instruments:

Internation Trauma Questionnaire (ITQ). Based on the ICD-11 criteria for diagnosing PTSD and complex PTSD, the ITQ(4) assesses both, symptoms and functional impairment in the past month. Six items measure core elements of PTSD (reexperiencing, avoidance and sense of threat), and an additional six items measure three

aspects of disturbances in self-organization, a core element of CPTSD (affective dysregulation, negative self-concept and disturbances in relationships). Both symptom assessments are followed by three questions about whether the symptoms have affected different areas of life. All 18 items are answered on a 5-point Likert scale from "not at all" to "extremely". In addition, subjects give a brief description of the traumatic event they experienced and indicate how long ago it occurred.

**Shutdown Dissociation Scale (Shut-D).** The Shut-D(7) measures three types of dissociation that can occur in PTSD: intrusion, hyperarousal and dissociation. The 13 items are evaluated based on experiences, on a 4-point Likert scale ranging from "not at all" to "5 or more times a week".

**Patient Health Questionnaire (PHQ-9).** The PHQ-9(3) is a brief questionnaire measuring nine symptoms of depression on a 4-point Likert scale from "not at all" to "almost every day". An additional question about the symptoms' effects on different areas of life is also rated on a 4-point Likert scale.

**Life Events Checklist (LEC-5).** The LEC-5 (6) measures life-time exposure to 17 categories of potentially traumatic events, including experiences with war, death, injury and assault. For each event category, different types of exposure are assessed: Happened to me, Witnessed it, Learned about it, Part of my job, Not sure, Doesn't apply.

#### Method:

The study will collect qualitative data in the form of participants' narratives that are created during the therapy sessions, and quantitative data in the form of questionnaires. For the treatment group, quantitative data will be collected at three timepoints: 1) a baseline screening measurement before treatment starts, 2) a post-treatment screening measurement after the last treatment session, and 3) a follow-up screening measurement six months after treatment completion. For the control group, data will be collected at baseline and post-treatment (i.e. after the waiting period that corresponds to the treatment group's treatment period). At each timepoint, the following instruments will be used: Internation Trauma Questionnaire (ITQ) (4)an 18-item questionnaire measuring elements of PTSD and complex PTSD as well as functional impairment; the Shutdown Dissociation Scale (Shut-D) (7), measuring three types of dissociation in PTSD; and the Patient Health Questionnaire (PHQ-9) (10) measuring nine symptoms of depression as well as functional impairment. At baseline, participants will also fill in the Life Events Checklist (LEC-5) (6), measuring different types of exposure to 17 categories of potentially traumatic events. In addition, demographic data, including time in Norway, gender, age, marital status, highest level of education, long term illness, general view about the health, will be collected.

To investigate the effects of NET, linear mixed-effects models with fixed effects for Group (treatment, control) and Time (baseline, post-treatment, follow-up) and their interaction

(Group X Time) will be calculated for each of the three symptom measures; ITQ, Shut-D and PHQ-9. To investigate the effect of NET, a 2x2 ANOVA (between-subject factor group: treatment, control; within-subject factor timepoint: baseline, post-treatment) will be calculated for each of the three symptom measures, ITQ, Shut-D and PHQ-9. In order to investigate the long-term effects of NET and the development of symptoms over a longer time period, a Repeated Measures ANOVA will be calculated for the treatment group for baseline, post-treatment and follow-up assessments. Additional analyses will be calculated to investigate the effect of trauma exposure on baseline symptom severity, and the effect of baseline symptom severity on treatment effect/symptom reduction.

#### **Primary hypotheses:**

H1: Participants receiving NET will show a significantly greater reduction in PTSD symptoms (ITQ) from baseline to post-treatment than participants in the control group

H2: Participants receiving NET will show a significantly greater reduction in dissociation symptoms (Shut-D) from baseline to post-treatment than participants in the control group.

H3: Participants receiving NET will show a significantly greater reduction in depression symptoms (PHQ-9) from baseline to post-treatment than participants in the control group.

H4: Participants receiving NET will have significantly lower PTSD symptoms (ITQ) at sixmonths follow-up compared to baseline, with no significant differences between follow-up and post-treatment.

H5: Participants receiving NET will have significantly lower dissociation symptoms (Shut-D) at six-months follow-up compared to baseline, with no significant differences between follow-up and post-treatment.

H6: Participants receiving NET will have significantly lower depression symptoms (PHQ-9) at six-months follow-up compared to baseline, with no significant differences between follow-up and post-treatment.

## Secondary hypotheses:

H7: Direct Experience with the Event (Happened to me - LEC-5) will be associated with greater baseline symptom severity (ITQ, Shut-D, PHQ-9).

H8: Participants with greater baseline symptom severity will experience a greater reduction in symptoms from baseline to post-treatment, compared to participants with milder initial symptom severity.

H9: Change in narrative coherence mediates the reduction in PTSD symptoms from baseline to post-treatment.

#### **Embedded Qualitative Study:**

A qualitative substudy will be conducted alongside the RCT to explore participants' lived experiences of NET. This substudy will involve phronetic iterative thematic analysis(11) of anonymized therapy narratives collected during NET sessions. The analysis will alternate between inductive (emic) insights and theoretical (etic) interpretations to uncover how participants construct meaning from traumatic events, how narrative coherence evolves throughout therapy, and how identity reconstruction occurs post-trauma.

#### **Research Questions**

- How do Ukrainian refugees make sense of war-related trauma through narrative?
- What are the common thematic shifts in personal narratives before and after NFT?
- How is narrative coherence associated with psychological recovery?

#### Analytical Procedure (Step-by-Step)

- 1. **Data Organization**: Anonymized narratives are digitized and categorized by case and treatment stage (pre/post).
- 2. **Immersion**: Researchers read and reread the data, noting key emotional, temporal, and identity-related elements.
- 3. **Primary-Cycle Coding**: Open descriptive coding is conducted using NVivo, with in vivo labels capturing participant language and early conceptual codes.
- 4. **Codebook Development**: A preliminary codebook is created, refined after intercoder dialogue, including definitions, inclusion/exclusion criteria, and examples.
- 5. **Secondary-Cycle Coding**: First-level codes are clustered into second-level interpretive themes. Existing theoretical frameworks (e.g., NET theory, trauma recovery models) are used to deepen understanding.
- 6. **Thematic Mapping**: Themes are hierarchically organized to show narrative transformation (e.g., victimhood → resilience).
- 7. **Memo Writing**: Reflective analytic memos are produced iteratively to document insights and guide interpretation.
- 8. **Saturation and Triangulation**: Data is revisited until thematic saturation is achieved. Therapist notes and supervision feedback are triangulated to validate interpretations.

- 9. **Negative Case Analysis**: Deviant narratives are explored to refine and challenge emerging findings.
- 10. **Reporting**: Themes are described with illustrative quotes, connecting them to the guiding research questions and literature.

#### **Outcome Measures:**

#### **Primary Outcome Measures**

#### 1. PTSD Symptom Severity (ITQ)

- o Instrument: International Trauma Questionnaire (ITQ)
- Description: Assesses symptoms of PTSD and Complex PTSD, including re-experiencing, avoidance, threat perception, and functional impairment.
- o Time Points: Baseline, Post-treatment, 6-month Follow-up
- o Outcome Focus: Change in PTSD symptom scores over time (H1, H4)

#### 2. Dissociation Symptoms (Shut-D)

- o Instrument: Shutdown Dissociation Scale (Shut-D)
- Description: Measures dissociative responses specific to trauma, including cognitive-emotional shutdown, sensory-motor dissociation, and behavioral shutdown.
- o Time Points: Baseline, Post-treatment, 6-month Follow-up
- Outcome Focus: Change in dissociation symptom scores over time (H2, H5)

## 3. Depression Symptoms (PHQ-9)

- o Instrument: Patient Health Questionnaire-9 (PHQ-9)
- Description: Measures the frequency of depressive symptoms over the past two weeks, including somatic and cognitive-affective dimensions, plus functional impairment.
- o Time Points: Baseline, Post-treatment, 6-month Follow-up
- Outcome Focus: Change in depressive symptoms (H3, H6)

#### **Secondary Outcome Measures**

## 4. Exposure to Traumatic Events (LEC-5)

o Instrument: Life Events Checklist for DSM-5 (LEC-5)

- Description: Captures direct and indirect exposure to 17 categories of potentially traumatic events, including whether the event "happened to me."
- Time Point: Baseline
- Outcome Focus: Association between level of trauma exposure and symptom severity (H7)

#### 5. Narrative Coherence (Qualitative Coding)

- Instrument: Qualitative content analysis or validated narrative coherence scale (to be specified in analytic plan)
- Description: Evaluates improvement in the structure, clarity, and emotional processing of the autobiographical trauma narrative as constructed during NET.
- $\circ$  Time Points: Session 2 (Lifeline) vs Session 7 (final exposure)
- Outcome Focus: Mediation analysis of change in PTSD symptoms through increased narrative coherence (H9)

## **Other Pre-Specified Measures**

#### 7. Demographic Variables

- o Instrument: Custom questionnaire
- o Description: Age, gender, marital status, education, time in Norway, long-term illness, and general health perception
- o Time Point: Baseline
- o Analytical Use: Covariates or moderators in outcome models

# 8. Functional Impairment

- o Embedded in: ITQ and PHQ-9
- o Description: Assesses impact of PTSD and depression on daily functioning
- $\circ \quad \textit{Time Points: } \textbf{Baseline, Post-treatment, 6-month Follow-up}$
- o Outcome Focus: Supplementary analysis of clinical relevance

## References:

- 1. UNHCR. The Operational Data Portal 2025 [cited 2025 22.05]. UNHCR webpage ]. Available from: https://data.unhcr.org/en/situations/ukraine.
- 2. Schauer M, Neuner F, Elbert T. Narrative Exposure Therapy (NET) For Survivors of Traumatic Stress. 3 ed: Hogrefe Publishing; 2025.
- 3. Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001;16(9):606-13.
- 4. Cloitre M, Shevlin M, Brewin C, Bisson J, Roberts N, Maercker A, et al. International trauma questionnaire. European Journal of Trauma & Dissociation. 2018.
- 5. Gray MJ, Litz BT, Hsu JL, Lombardo TW. Psychometric properties of the life events checklist. Assessment. 2004;11(4):330-41.
- 6. Weathers FW, Blake, D.D., Schnurr, P.P., Kaloupek, D.G., Marx, B.P., & Keane, T.M. The Life Events Checklist for DSM-5 (LEC-5) 2013 [Available from: <a href="https://www.ptsd.va.gov">www.ptsd.va.gov</a>.
- 7. Schalinski I, Maggie S, and Elbert T. The Shutdown Dissociation Scale (Shut-D). European Journal of Psychotraumatology. 2015;6(1):25652.
- 8. Labberton AS, Ozeryansky L, Helland Y, Skogheim TS, Hansen TM. Trends in the health status of Ukrainian refugees in Norway according to month of arrival during 2022. BMC Public Health. 2024;24(1):3127.
- 9. Labberton AS, Hansen TM, Skogheim TS, Helland Y. Healthcare needs among refugees from Ukraine arriving in Norway during 2022. Norwegian Institute of Public Health; 2023 May 2023.
- 10. Ardino V, Schalinski I. Recent developments of narrative exposure therapy. Maltrattamento e Abuso All'Infanzia: Rivista Interdisciplinare. 2020;.22(3):pp.
- 11. Tracy SJ. A phronetic iterative approach to data analysis in qualitative research. 질적연구. 2018;19(2):61-76.